CLINICAL TRIAL: NCT01301703
Title: The Efficacy and Safety of Vaccination Against Pertussis. Tetanus and Diphtheria in Patients Suffering From Rheumatoid Arthritis
Brief Title: Vaccination Against Pertussis, Tetanus and Diphtheria in Patients Suffering From Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Ori Elkayam, Department of Rheumatology. Tel Aviv Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0068-09
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid pertussis tetanus
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tdap vaccination (Active Comparator): Patients and controls will be vaccinated with BOOSTRIX (Tdap vaccine)
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine, Adsorbed)

INTERVENTIONS:
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine, Adsorbed) — a single 0.5-mL intramuscular injection into the deltoid muscle of the upper arm

SUMMARY:
Pertussis is an acute respiratory infection caused by Bordetella pertussis. Rates of recent B. pertussis infection between 8%--26% have been reported among adults with cough illness of at least 5 days duration who sought medical care. The CDC recommends vaccinating patients aged 15 to 64 years old, once in 10 years. Although acellular vaccines such as BOOSTRIX have been evaluated in healthy population, the safety and efficacy of this vaccine in patients suffering from rheumatic diseases have not been established.

Study population : 50 Rheumatoid Arthritis (RA) patients and 5 healthy controls

Evaluation : the evaluation will be performed on week 0 and 4-6 weeks later. In terms of safety, the patients will be evaluated according to the Disease Activity Index (DAS). Blood will be drawn at each visit at tested for humoral response to tetanus and pertussis.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from RA
* Aged 18 to 64 years old

Exclusion Criteria:

* Active disease requiring a change in drug regimen
* Known allergy to vaccine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of Tdap in patients suffering from rheumatoid arthritis | 4-6 weeks after vaccination
  Geometric mean titers and individual responses to components of pertussis, tetanus and diphtheria

SECONDARY OUTCOMES:
Safety of Tdap vaccine in RA patients | 4-6 weeks after vaccination
  Safety will be evaluated using the disease activity score (DAS) at baseline and 4-6 weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Tel Aviv Medical Center, Tel Aviv, Israel